CLINICAL TRIAL: NCT07166341
Title: Accuracy Performance Verification of the INVOS™ PM7100 System, Comparing rSO2 Values to Reference Blood Oxygen Saturation Measurements in Adult Human Volunteers
Brief Title: Accuracy Verification of the INVOS PM7100
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT24046IN4WVL
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Tissue Oxygenation
Keywords: NIRS, INVOS, Tissue Oxygenation, Regional Oxygenation
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy, non-smoking volunteers ages ≥18 to <47 years who meet inclusion criteria
  Interventions: Device: Observational

INTERVENTIONS:
Device: Observational — The study objectives require placement of a jugular venous bulb catheter and radial arterial line placement with ultrasound guidance. Two INVOS™ sensors (PMSENS71-A) will be placed bilaterally on the subject's forehead and two on the calf. The INVOS™ device will be evaluated for a targeted range of 70-100% SpO2 levels. Hypoxic mixtures of gas are delivered, and data are collected at approximately (~) 5-minute intervals during steady periods of increasing and decreasing oxygen concentration.

SUMMARY:
Prospective, observational, pre-market, verification study to confirm accuracy of the INVOS 7100 system in compliance with ISO 80601-2-85:2021 standard

DETAILED DESCRIPTION:
Verify that the INVOS PM7100 system in conjunction with the INVOS Adult Sensors meets the requirements for tissue saturation accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of ≥18 to <47 years
* Completion of a health screening for medical history by a licensed physician, nurse practitioner, or physician assistant
* Subject is a non-smoker or has not smoked within 2 days prior to the study
* Minimum weight 40kg
* BMI within range 18.0-- 35.0
* Reference tissue hemoglobin oxygen saturation over the range 50% to 85%

Exclusion Criteria:

* Compromised circulation, injury, or physical malformation of fingers, hands, or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study (Note: certain malformations may still allow subjects to participate if the condition is noted and would not affect the sites utilized)
* Prior or known allergies to lidocaine (or similar pharmacologic agents, e.g., Novocain) [self-reported]
* Prior known severe allergies to medical grade adhesive/tape (Band-Aid) [self-reported]
* Subjects taking certain medication(s) beyond birth control may be excluded from participating at the PI discretion [self-reported]
* Subject participation will be at the PI's discretion if they are currently participating in, or if they have recently participated in (discontinued within 30 days prior to the hypoxia procedure for this study) in an investigational drug, device, or biologic study [self-reported]
* Negative Allen's test for radial and ulnar patency
* Has made a whole blood donation or has had at least 450 ml of blood drawn within 8 weeks prior to the study procedure [self-reported]
* Individuals of childbearing potential who are pregnant, who are trying to get pregnant, or who have a urine test positive for pregnancy on the day of the study and is unwilling to use effective birth control between the time of screening and study procedure, or is breastfeeding.
* Has anemia [lab values specific for gender]
* Has a history of sickle cell trait or thalassemia [self-reported]
* Has an abnormal hemoglobin electrophoresis test [lab measurement]
* Has a positive urine cotinine test or urine drug screen or oral ethanol test [Point of Care (POC) testing]
* Has a room air saturation less than 95% by pulse oximetry [measurement by PI or delegate]
* Has a clinically significant abnormal ECG [assessment by PI or delegate]
* Has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate]
* Has a COHb greater than 3%, or MetHb greater than 2% [measured by venous blood sample co-oximetry]
* Has tHb < 10 g/dl as assessed by co-oximetry during the procedure

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, non-smoking volunteers ages of ≥18 to <47 years who meet inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Accuracy in terms of the root mean square error | Performance evaluation is expected take approximately 2.5 hours
  Performance assessed by comparing INVOS™ rSO2 to the calculated global field saturation (fSO2) value obtained from simultaneous arterial and jugular venous blood samples during normocapnia.

SECONDARY OUTCOMES:
Trend accuracy | Evaluation is expected take approximately 2.5 hours
  * Cerebral site: Complete system in conjunction with an adult sensor (model PMSENS71-A) shall have an rSO2 trending accuracy over the declared range of 50% to 85% compared to reference hemoglobin tissue oxygen saturation.
  * Somatic site: System shall be able to calculate rSO2 on somatic sites.
Trend accuracy in a hypercapneic state | Evaluation is expected take approximately 2.5 hours
  Device performance will be evaluated during hypercapnia

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, MDDS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States